CLINICAL TRIAL: NCT04845945
Title: Response to Guideline-concordant Pneumococcal Vaccination Strategy in Cardiac Transplant Candidates and Recipients
Brief Title: MISP 60528 Pneumococcal Vaccination
Status: Terminated | Type: Observational
Why Stopped: Termination of funding by the sponsor/funder.
Sponsor: Montefiore Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Sunfire Biotechnologies (Unknown); Quest Clinical Research (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-12637; MISP 60528 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2021-03-19; First posted 2021-04-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Heart Transplant Infection Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PCV15 only: Draw blood for ELISA and OPA, then administer PCV15
  Interventions: Biological: PCV15
- PPS23 only: Draw blood for ELISA and OPA, then administer PPS23
- PCV15 and PPS23: Draw blood for Administer PPS23 then draw blood again ELISA and OPA, then administer PCV15
  Interventions: Biological: PCV15

INTERVENTIONS:
Biological: PCV15 — Blood draw after the vaccination
  Other Names: PPS23; PCV15 and PPS23
  Groups: PCV15 and PPS23; PCV15 only

SUMMARY:
This study aims to use two different blood tests (ELISA and OPA) to study response to pneumococcal vaccination administered as per standard guidelines in patients who are undergoing workup for heart transplant (whether or not they have undergone LVAD implantation or have undergone heart transplant.

DETAILED DESCRIPTION:
The patients will be receiving vaccination consistent with standard of care guidelines, regardless of study participation. The additional risk of study participation would be the risks associated with venipuncture (injury to vessel or nerve, syncope).

Patients will not accrue benefits personally. However, participation will help others by identifying whether current vaccination strategies in this population are adequate.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Either undergoing evaluation for heart transplant (with or without LVAD receipt), or having received a heart transplant
* Receiving a dose of PCV15 or PPSV23 (or both sequentially) concordant with AST guidelines

Exclusion Criteria:

* Infants and children under age 18
* Subjects without the capacity to consent
* Pregnancy
* Already up to date on pneumococcal vaccination or declining vaccination

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We are excluding infants and children as they are immunologically different from adults, respond to vaccinations differently, and guidelines for childhood vaccination are different from those for adult vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-08-24 (Actual)

PRIMARY OUTCOMES:
Vaccine response | 12 weeks
  Antibody levels

SECONDARY OUTCOMES:
Serotype ELISA response | 12 weeks
  Antibody production to specific serotype

CONTACTS AND LOCATIONS:
Overall Officials: Vagish Hemmige, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, Infectious Diseases, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No